CLINICAL TRIAL: NCT06053268
Title: Mindfulness Interventions to Improve Health Activation, Coping, and Stress Among Childhood Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MINDHACS; NCI-2023-09351 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2023-09-07; First posted 2023-09-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Leukemia; Lymphoma; Childhood Cancer
MeSH Terms: conditions — Leukemia; Lymphoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single-arm, within-subject pilot: EmbracePlus smartwatch (Experimental): Prior to engaging in the intervention participants will complete baseline assessments of stress and coping. Participants will then engage in a daily mindfulness practice via the Headspace mobile application. The basic application program includes daily 10-minute sessions in guided mindfulness meditation that include mindful breathing, body awareness, emotion and thought recognition, and attentional control. During the first and fourth week of the intervention, participants will complete EMAs assessing mood, current activity, and intervention engagement. Participants will also wear a wrist-worn device to assess biomarkers of stress. At the completion of the intervention participants will complete follow-up assessments related to intervention and data collection procedures feasibility and acceptability as well as coping behaviors and stress.
  Interventions: Device: Headspace

INTERVENTIONS:
Device: Headspace — The intervention will be delivered via the Headspace mobile application. The basic application program includes daily 10-minute sessions in guided mindfulness meditation that include mindful breathing, body awareness, emotion and thought recognition, and attentional control

SUMMARY:
This study will explore feasibility and acceptability of using a daily mobile mindfulness app to cope with stress. In addition, feasibility of digital health data collection procedures including wrist-worn devices and ecological momentary assessments will be examined.

PRIMARY OBJECTIVES

* Determine the feasibility and acceptability of completing the 30-day mobile mindfulness program
* Evaluate the feasibility of digital health data collection procedures to detect autonomic nervous system (ANS) activation associated with stress (e.g., electrodermal activity, pulse rate variability, skin temperature) via wearable devices and self-reported ecological momentary assessments (EMA) among adult survivors of childhood cancer in the SJLIFE cohort
* Generate preliminary data to estimate the effect size and power needed for an extramurally funded randomized controlled trials (RCT) examining the impact of daily mindfulness mediation on biomarkers of ANS activation, coping, health behaviors, and cardiometabolic outcomes in a cohort of survivors of childhood cancer.

DETAILED DESCRIPTION:
Prior to engaging in the intervention participants will complete baseline assessments of stress and coping. Participants will then engage in a daily mindfulness practice via the Headspace mobile application. The basic application program includes daily 10-minute sessions in guided mindfulness meditation that include mindful breathing, body awareness, emotion and thought recognition, and attentional control. During the first and fourth week of the intervention, participants will complete EMAs assessing mood, current activity, and intervention engagement. Participants will also wear a wrist-worn device to assess biomarkers of stress. At the completion of the intervention participants will complete follow-up assessments related to intervention and data collection procedures feasibility and acceptability as well as coping behaviors and stress.

ELIGIBILITY:
Inclusion Criteria:

* Research participant is at least 18 years old at enrollment
* Research participant is followed by St. Jude Children's Research Hospital (SJCRH)
* Research participant has a diagnosis history of leukemia or lymphoma
* Research participant takes part in the St. Jude Lifetime Cohort Study (SJLIFE)
* Research participant has elevated psychological stress scores of 6 or greater on most recent SJLIFE questionnaire
* Participant can speak and read English

Exclusion Criteria:

* Research participant currently engages in mindful stress-reduction practices >2x per week (e.g., tai chi, meditation)
* Research participant takes psychiatric medications or medications that impact cardiac functioning, beta-blockers, alpha-blockers
* Research participant wears a pacemaker
* Research participant has a diagnosis of a congenital heart disease
* Research participant has no access to a smartphone
* Research participant has elevated pain interference scores (T≥70)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2026-09-27 (Estimated)

PRIMARY OUTCOMES:
Intervention feasibility. | 30 days (during intervention
  Headspace provides user metrics including date/time of meditation sessions, number of sessions completed, average duration of each session, and total meditation minutes overall.
Intervention acceptability | up to 1 week post intervention]
  Treatment Acceptability and Adherence Scale- Participants will rate on a 0 ("Strongly disagree") to 7 ("Strongly agree") scale regarding their perceptions of acceptability of the mindfulness intervention (10 items).
Data collection feasibility. | up to 1 week post intervention
  Wearable Technology. EmbracePlus includes on-wrist detection, and this data will be used to evaluate how long and for how many days participants wear the device.
  EMA. Completion of EMA data will be calculated based on the number of assessments completed
EMA data collection acceptability | up to 1 week post intervention
  An adapted version of the TAAS was created to evaluate EMA assessment acceptability (7 items). Higher scores are indicative of greater acceptability

SECONDARY OUTCOMES:
Perceived Stress Scale | Baseline and up to 1 week post intervention
  This measure is a 10-item, widely used and validated assessment of stress and efficacy of managing stress. The Participants are asked to respond to each question on a 5-point Likert scale ranging from 0 (never) to 4 (very often), indicating how often they have felt or thought a certain way within the past month. Scores range from 0 to 40.
Brief Cope inventory is a 28-item, validated assessment measure of positive and negative coping strategies across 14 domains. Participants respond on a 4 point Likert scale how often they have engaged in a particular coping strategy | Baseline and up to 1 week post intervention
  Digital biomarkers of ANS activation. EmbracePlus (Empatica, Milano, Italy) is a smartwatch engineered to collect physiological biomarkers associated with ANS activation including electrodermal activity (EDA), pulse rate variability, inter-beat interval, respiratory rate, skin temperature, blood volume pulse- each used to develop a stress experience composite score

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Webster, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols